CLINICAL TRIAL: NCT01471626
Title: Real-time Attended Home-polysomnography Through Telematic Data Transmission
Acronym: sleepbox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, pneumologist, chef de clinique adjoint, Centre Hospitalier Universitaire Saint Pierre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK/-10-81/4077
Record Dates: First submitted 2011-10-10; First posted 2011-11-15 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; polysomnography; telemedicine
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- telematic attended polysomnography (Experimental)
  Interventions: Device: polysomnograph Dream and Sleep Box

INTERVENTIONS:
Device: polysomnograph Dream and Sleep Box — Portable polysomnograph will be placed at home around 7:00PM. The Sleep Box (wireless monitoring device) will be left near the patient, to allow real-time GPRS transmission of recorded sleep parameters to the sleep lab.

SUMMARY:
The purpose of this study is to develop an efficient home-based polysomnography device, which allows, through GPRS,continuous real-time monitoring from the sleep lab based in the hospital, in order to decrease the failure rate of home-based recordings.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of OSA
* 18 y old

Exclusion Criteria:

* restrictive respiratory disorders
* distance home-hospital exceeding 30 Km.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Principal Investigator — CHU St Pierre
Locations (1):
- CHU St Pierre, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in the Sleep Lab of a tertiary hospital. Patients were recruted for ploysomnography if they were clinically suspicted of OSA.
Groups:
- Telematic Attended Polysomnography: All patients underwent one Home-PSG, using Dream and Sleepbox (Medatec, Belgium), that is a wireless system able to communicate with Dream, and with Internet through a wi-fi/3G interface. It is equipped with a digital infrared camera, and with a speaker/microphone system for bidirectional audio/video communication via Skype.
  The Sleep Lab nurse performed a discontinue monitoring of the PSG. In case of defective signals, she called the patient who had been previously educated to replace the sensors.
Period: Overall Study
Arm/Group | Telematic Attended Polysomnography
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Telematic Attended Polysomnography
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  Belgium | 21

OUTCOME MEASURES:

1. Primary Outcome: Quality of Polysomnographic Recordings
Description: Quality of recordings will be graded according to Redline S et al (SLEEP 1998): Unsatisfactory, poor, fair, good, very good,excellent. Unsatisfactory and poor recordings are considered as failures.
Time Frame: 1 week
Measure: Number; unit: percentage of recording failure
Arm/Group | Telematic Attended Polysomnography
Number analyzed (Participants) | 21
percentage of recording failure | 10

ADVERSE EVENTS:
Arm/Group | Telematic Attended Polysomnography
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
-technical problems with the Skype® connection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No